CLINICAL TRIAL: NCT00665847
Title: A Phase II, Open-label Trial, to Evaluate the Safety, Tolerability and Antiviral Activity of TMC125 in Antiretroviral Experienced HIV-1 Infected Children and Adolescents
Brief Title: TMC125-TiDP35-C213: Safety and Antiviral Activity of Etravirine (TMC125) in Treatment-Experienced, HIV Infected Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002746; TMC125-TiDP35-C213 (Other: Tibotec Pharmaceuticals, Ireland); 2007-007086-21 (EudraCT Number); NCT00750542 (obsolete NCT alias)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: HIV-1
Keywords: HIV-1; TMC125-TiDP35-C213; TMC125-C213
MeSH Terms: interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etravirine (TMC125) (Experimental)
  Interventions: Drug: Etravirine (TMC125); Drug: Optimized background regimen (OBR)

INTERVENTIONS:
Drug: Etravirine (TMC125) — Patients will be dosed by body weight , i.e. 5.2 mg/kg twice daily (b.i.d.) up to a maximum of 200 mg b.i.d. for 48 weeks.
Drug: Optimized background regimen (OBR) — An investigator-selected optimized background regimen (OBR) comprising of a low-dose ritonavir (rtv)-boosted protease inhibitor (PI) (either lopinavir [LPV], darunavir [DRV], atazanavir [ATV] or saquinavir [SQV]) in combination with nucleos(t)ide reverse transcriptase inhibitor(s) (N[t]RTIs) to be dosed according to the drugs individual package inserts for 48 weeks.

SUMMARY:
The purpose of this study is to determine the safety and antiviral activity of etravirine in treatment-experienced human immunodeficiency virus (HIV) infected children and adolescents.

DETAILED DESCRIPTION:
The study design is a single arm treatment (all patients assigned to receive etravirine), open label (patients will know the identity of the treatments they are receiving) safety and antiviral activity of Etravirine (TMC125) in treatment-experienced, HIV infected children and adolescents 6 to 17 years of age. Etravirine is a new drug belonging to the NNRTI (a non-nucleoside reverse transcriptase inhibitor) drug class that slows down the growth of the human immunodeficiency virus (HIV). This drug has been tested for safety and effectiveness in adults, however, there is no data on the drug's long-term safety and antiviral activity in children and adolescents. This study will last for a maximum of 48 weeks. A total of 100 ptients will receive etravirine tablets based on body weight and an investigator selected optimized background regimen (OBR) of at least 2 antiretrovirals (ARVs), consisting of a boosted protease inhibitor (PI) and nucleoside reverse transcriptase inhibitor(s) (NRTI[s]). Use of enfuvirtide is optional. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Body weight according to age within the 10-90th percentile of CDC growth chart
* On steady antiretroviral therapy regimen for at least 8 weeks at screening and willing to remain on that regimen until baseline
* HIV viral load of 1,000 copies/ml or greater at study entry
* Parent or legal guardian willing to provide informed consent, if necessary

Exclusion Criteria:

* The Key Exclusion Criteria are: Evidence of resistance to etravirinel Any grade 3 or 4 toxicity (More information available in the protocol)
* Use of disallowed concomitant therapy (specified in the protocol)
* Currently active AIDS defining illness (category C)
* Active hepatitis A, B or C virus infection
* Any clinically significant diseases or findings that, in the opinion of the investigator, would interfere with the study
* Receipt of any ARV or non-ARV investigational medication or investigational vaccine within 30 days prior to screening
* History of clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication (TMC125)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2008-11; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (42):
- United States (13):
  - Mobile, Alabama
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - New Orleans, Louisiana
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - New York, New York
  - Syracuse, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
- Buenos Aires, Argentina
- Brazil (3):
  - Belo Horizonte
  - Ribeirão Preto
  - Rio de Janeiro
- Canada (3):
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (4):
  - Lyon
  - Nantes
  - Paris
  - Toulouse Cedex 3 N/A
- Amsterdam-Zuidoost, Netherlands
- Portugal (3):
  - Almada
  - Lisbon
  - Porto
- Puerto Rico (2):
  - Rio Piedras
  - San Juan
- Romania (2):
  - Bucharest
  - Constanța
- South Africa (3):
  - Dundee
  - Durban
  - Port Elizabeth
- Spain (4):
  - Barcelona
  - Esplugues de Llobregat
  - Madrid
  - Seville
- Thailand (2):
  - Bangkok
  - Khon Kaen
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Tambuyzer L, Thys K, Hoogstoel A, Nijs S, Tomaka F, Opsomer M, De Meyer S, Vingerhoets J. Assessment of etravirine resistance in HIV-1-infected paediatric patients using population and deep sequencing: final results of the PIANO study. Antivir Ther. 2016;21(4):317-27. doi: 10.3851/IMP3011. Epub 2015 Nov 13. PMID 26566161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 41 investigators in 13 countries enrolled patients in study TMC125-C213. A total of 103 patients were documented as being enrolled in the study, however 2 patients were randomized in error. Therefore, 101 patients were enrolled and treated with etravirine (ETR) also known as TMC125 and included in the intent-to-treat (ITT) population.
Groups:
- TMC125: TMC125 dosed according to body weight (kg) from 100 mg to 200 mg twice a day
Period: Overall Study
Arm/Group | TMC125
Started | 101
Completed | 76
Not Completed | 25
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 2
Not completed — Subject non-compliant | 8
Not completed — Subject reached a virologic endpoint | 4
Not completed — Resistance to TMC125 | 1
Not completed — Subject ineligible to continue the trial | 1
Not completed — Switch to Commercial Medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | TMC125
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (2.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 37
Age Customized [Number; unit: participants]
  >=6 to <12 years | 41
  >=12 to <18 years | 60

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) was defined as an event that occurred in the 48-week treatment period during which it emerged (i.e. started or worsened in severity, relation, or other attribute), and not in the subsequent study periods, even if the event continued to be present. Adverse events were graded from 1 to 4 in severity using the Division of Acquired Immunodeficiency Syndrome severity scale (grade 1 being less severe and grade 4 being more severe). ETR=etravirine/TMC125; OBR=optimized background regimen
Time Frame: 48 weeks
Population: The safety analysis was done on the intent-to-treat (ITT) population, which included all patients who received at least one dose of investigational medication.
Measure: Number; unit: Patients
Groups:
- TMC125: TMC125 dosed based on body weight (kg) from 100 mg to 200 mg twice a day
Arm/Group | TMC125
Number analyzed (Participants) | 101
Patients
  Any TEAE | 89
  TEAEs that were fatal | 0
  TEAEs that were serious | 5
  TEAEs that were grade 3 or 4 in severity | 14
  TEAEs leading to temporary ETR discontinuation | 8
  TEAEs leading to permanent ETR discontinuation | 8
  TEAEs possibly related to ETR | 23
  TEAEs probably related to ETR | 14
  TEAEs very likely related to ETR | 3
  TEAEs at least possibly related to ETR | 33
  TEAEs possibly related to OBR | 27
  TEAEs probably related to OBR | 12
  TEAEs very likely related to OBR | 5
  TEAEs at least possibly related to OBR | 36
  TEAEs of at least grade 2 in severity | 21
  TEAEs of at least grade 3 in severity | 3
  TEAEs of interest: Skin event | 31
  TEAEs of interest: Rash | 23
  TEAEs of interest: severe cutaneous reactions | 7
  TEAEs of interest: angioedema | 4
  TEAEs of interest: neuropsychiatric events | 2
  TEAEs of interest: hepatic events | 0
  TEAEs of interest: cardiac events | 0
  TEAEs of interest: bleeding events | 0
  TEAEs of interest: pancreatic events | 1
  TEAEs of interest: lipid-related events | 6
  TEAEs of interest: neoplasms | 1

2. Primary Outcome: The Percentage of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: The percentage of patients with a treatment-emergent adverse event (TEAE) (defined as an event that occurred in the 48-week treatment period during which it emerged [i.e. started or worsened in severity, relation, or other attribute], and not in the subsequent study periods, even if the event continued to be present] are provided below. Adverse events were graded from 1 to 4 in severity using the Division of Acquired Immunodeficiency Syndrome severity scale (grade 1 being less severe and grade 4 being more severe). ETR=etravirine/TMC125; OBR=optimized background regimen
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | TMC125
Number analyzed (Participants) | 101
Percentage of patients
  Any TEAE | 88.1
  TEAEs that were fatal | 0
  TEAEs that were serious | 5.0
  TEAEs that were grade 3 or 4 in severity | 13.9
  TEAEs leading to temporary ETR discontinuation | 7.9
  TEAEs leading to permanent ETR discontinuation | 7.9
  TEAEs possibly related to ETR | 22.8
  TEAEs probably related to ETR | 13.9
  TEAEs very likely related to ETR | 3.0
  TEAEs at least possibly related to ETR | 32.7
  TEAEs possibly related to OBR | 26.7
  TEAEs probably related to OBR | 11.9
  TEAEs very likely related to OBR | 5.0
  TEAEs at least possibly related to OBR | 35.6
  TEAEs of at least grade 2 in severity | 20.8
  TEAEs of at least grade 3 in severity | 3.0
  TEAEs of interest: Skin event | 30.7
  TEAEs of interest: Rash | 22.8
  TEAEs of interest: severe cutaneous reactions | 6.9
  TEAEs of interest: angioedema | 4.0
  TEAEs of interest: neuropsychiatric events | 2.0
  TEAEs of interest: hepatic events | 0
  TEAEs of interest: cardiac events | 0
  TEAEs of interest: bleeding events | 0
  TEAEs of interest: pancreatic events | 1.0
  TEAEs of interest: lipid-related events | 5.9
  TEAEs of interest: neoplasms | 1.0

3. Secondary Outcome: Population Pharmacokinetic (PK) Estimates of Etravirine/TMC125 (ETR): Area Under the Plasma Concentration-time Curve Over 12 Hours at Steady-state (AUC12h)
Description: The AUC12h is a Bayesian estimation based on a population pharmacokinetic model and sparse samples collected at each visit over the duration of trial. For each sparse sample taken, the time blood sample was recorded as well as the time of etravirine intake just prior to the time of blood sample.
Time Frame: Weeks 4-48
Population: The intent-to-treat (ITT) population, i.e. all patients who had been enrolled and taken ETR at least once, regardless of their compliance with the protocol was used for this analysis. The table below shows results for "Overall (children and adolescents combined)."
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | TMC125
Number analyzed (Participants) | 101
ng.h/mL | 5216 (4305)

4. Secondary Outcome: Population Pharmacokinetic (PK) Estimates of Etravirine/TMC125 (ETR): Trough Plasma Concentration (C0h)
Time Frame: Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC125
Number analyzed (Participants) | 101
ng/mL | 346 (342)

5. Secondary Outcome: Population Pharmacokinetic (PK) Estimates of Etravirine/TMC125 (ETR): Maximum Plasma Concentration (Cmax)
Description: Etravirine/TMC125 (ETR) Cmax was approximated for each individual using the median value of plasma ETR concentrations taken 4 hours postdose (± 1 hour), when available, on the day of the Week 4 visit as shown in the table below.
Time Frame: Week 4
Population: The intent-to-treat (ITT) population, i.e. all patients who had been enrolled and taken Etravirine/TMC125 (ETR) at least once, regardless of their compliance with the protocol was used for this analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC125
Number analyzed (Participants) | 101
ng/mL | 589 (486)

6. Secondary Outcome: Percentage of Patients With Virologic Response at Week 24
Description: Virologic response was defined as the percentage of patients with plasma viral load < 50 copies/mL at Week 24 calculated according to the non-completer=failure (NC=F) imputation method.
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of Patients
Arm/Group | TMC125
Number analyzed (Participants) | 101
Percentage of Patients | 52.5
Statistical Analysis 1: Comparison: TMC125; Test type: Superiority or Other; Proportion = 52.5, 95% CI 2-sided [42.7 to 62.2], Standard Error of Mean 0.050 — The standard error for a proportion was calculated as the square root of the variance divided by the number of patients. The variance for a proportion is equal to p*(1-p), with p being the proportion

7. Secondary Outcome: Change From Baseline in Human Immunodeficiency Virus - Type 1 (HIV-1) Ribonucleic Acid (RNA) in Plasma Over Time
Time Frame: Baseline, Week 48
Population: as for outcome 5
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | TMC125
Number analyzed (Participants) | 101
log10 copies/mL | -1.53 (0.132)

8. Secondary Outcome: The Change From Baseline in CD4 Cell Counts Over Time
Time Frame: Baseline, Week 48
Population: as for outcome 5
Measure: Mean (Standard Error); unit: 10E6 cells/L
Arm/Group | TMC125
Number analyzed (Participants) | 101
10E6 cells/L | 156 (22.7)

9. Secondary Outcome: The Emergence of Non-nucleoside Reverse Transcriptase Inhibitor Resistance-associated Mutations (NNRTI RAMs) in Patients Classified as Virologic Failures
Description: Virologic failure (lack of response) was defined as: plasma viral load decline of < 0.5 log10 from Baseline by Week 8 and/or plasma viral load decline of <1.0 log10 from Baseline by Week 12. Virologic failure (loss of response) was defined as 2 consecutive measurements of plasma viral load > 0.5 log10 above the nadir after a minimum of 12 weeks of treatment. The table below provides data for 41 viologic failures of which 30 had mutation data available. In the table below, only the 4 most frequently emerging mutations are presented (emerging in at least 3 patients).
Time Frame: Baseline and Endpoint (up to Week 48)
Population: The patients in the intent-to-treat (ITT) population classified as virologic failures were used for this analysis.
Measure: Number; unit: Patients
Arm/Group | TMC125
Number analyzed (Participants) | 41
Patients
  V90I | 3
  L100I | 3
  E138A | 3
  Y181C | 8

ADVERSE EVENTS:
Description: Only subjects who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. subjects with Non-Serious Adverse Events.
Arm/Group | TMC125
Serious Adverse Events (participants affected / at risk) | 5/101
Other Adverse Events (participants affected / at risk) | 70/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC125 (N=101)
Ulcerative keratitis (Eye disorders) | 1
Drug resistance (General disorders) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Immunoglobulins (Investigations) | 1
Lymphocyte morphology abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Treatment noncompliance (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC125 (N=101)
Conjunctivitis (Eye disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 11
Pyrexia (General disorders) | 9
Bronchitis (Infections and infestations) | 9
Oral herpes (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 8
Rhinitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 27
Headache (Nervous system disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less